CLINICAL TRIAL: NCT05526638
Title: Estimation of Serum and Tissue Level of Interleukin-15 (IL-15) and IL-15 Receptor Alpha (IL-15Rα) in Mycosis Fungoides Before and After Treatment
Brief Title: Serum and Tissue Level of Interleukin-15 (IL-15) and IL-15 Receptor Alpha (IL-15Rα) in Mycosis Fungoides
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mogawer, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MF-6-22
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New/ recurrent mycosis fungoides patients (Experimental): New' Recurrent mycosis fungoides treatment will receive be assessed for both serum and tissue levels of IL-15 and IL-15 Rα prior to and after treatment with phototherapy
  Interventions: Radiation: ultraviolet phototherapy

INTERVENTIONS:
Radiation: ultraviolet phototherapy — thrice weekly sessions of ultraviolet phototherapy

SUMMARY:
Estimation of serum and tissue level of IL-15 and IL-15 R α in mycosis fungoides prior to after treatment.

DETAILED DESCRIPTION:
Twenty patients will be recruited from the cutaneous lymphoma clinic who are either recently diagnosed with MF or presenting with recurrent MF following cessation of treatment.

An informed written consent will be obtained from all patients. Clinical assessment: Patients will be assessed clinically for extent by BSA as well as MF staging and type.

For MF staging, in addition to extent, diagnostic skin biopsies will be assessed for depth of the infiltrate. Radiological assessment including chest x-ray, pelvi-abdominal ultrasound as well as lymph node examination, ultrasound and biopsy if required. Biochemical assessment including complete blood count, liver and kidney function tests, lipid profile as well as lactate dehydrogenase and beta 2 microglobulin.

Standardized photographs will be taken at initial assessment as well as following resolution of the biopsied lesion.

Baseline biochemical assessment at the beginning of the study: Serum samples as well as 4mm lesional punch skin biopsies will be taken prior to starting phototherapy treatment to assess serum and tissue level of IL-15 and IL-15 R α level using enzyme-linked immunosorbent assay (ELISA).

Phototherapy treatment: Patients with superficial lymphocytic infiltrate will be assigned to either NB-UVB sessions, while those with deep infiltrate will be assigned to PUVA. Patients will undergo thrice weekly sessions.

Patients will be clinically assessed on monthly basis to monitor response to treatment and record any side effects.

Biochemical reassessment: Serum and lesional biopsies will be retaken following resolution of the biopsied lesion to assess serum and tissue level of IL-15 and IL-15 R α level using enzyme-linked immunosorbent assay (ELISA).

Afterwards, the biopsied lesion will be covered if the patients was having other unresolved lesions and monthly follow up will be carried to detect lesional recurrence. Any reported recurrence during the estimated study duration of 6 months will be re assessed for both serum and tissue level of IL-15 and IL-15 R α level using enzyme-linked immunosorbent assay (ELISA).

Twenty healthy controls will be recruited and assessed for both serum and tissue level of IL-15 and IL-15 R α level using enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mycosis fungoides; newly diagnosed or recurrent after cessation of treatment

Exclusion Criteria:

* Patients with any contraindication to phototherapy (e.g., any other skin cancers or photosensitivity); or to psoralen (e.g., liver disease).
* Subjects with history of solid or hematological malignancy as leukemia.
* Patients with autoimmune disease as SLE.
* Patients who received treatment for the past one month.
* Pregnant and lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessing percent change in serum and tissue levels of IL-15 and IL-15 Rα in cases of mycosis fungoides | 6 months
  Assessing percent change in serum and tissue levels of IL-15 and IL-15 Rα in cases of mycosis fungoides prior to starting phototherapy Assessing percent change in serum and tissue levels of IL-15 and IL-15 Rα in cases of mycosis fungoides prior to starting phototherapy and shortly after resolution of the biopsied lesion.
Assessing serum and tissue levels of IL-15 and IL-15 Rα in cases of mycosis fungoides prior to starting phototherapy in comparison to healthy controls. | 4 months
  Assessing serum and tissue levels of IL-15 and IL-15 Rα in cases of mycosis fungoides prior to starting phototherapy in comparison to healthy controls
Assessing serum and tissue levels of IL-15 and IL-15 Rα in cases of mycosis fungoides shortly after resolution of the biopsied lesion in comparison to healthy controls | 6 months
  Assessing serum and tissue levels of IL-15 and IL-15 Rα in cases of mycosis fungoides shortly after resolution of the biopsied lesion in comparison to healthy controls

SECONDARY OUTCOMES:
Feasibility of the use of serum levels of IL-15 and IL-15 Rα as markers for their tissue levels | 6 months
  Correlating serum level of serum levels of IL-15 and IL-15 Rα with their tissue levels

CONTACTS AND LOCATIONS:
Overall Officials: Randa Youssef, MD, Study Chair — Cairo University
Locations (1):
- Cutaneous Lymphoma clinic, Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participants' data that underlie reported results will be shared upon request, after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 12 months after article publication
Access Criteria: Controlled Access:
  Researchers who provide a methodologically sound proposal will be allowed to access data to achieve aims in the approved proposal.